CLINICAL TRIAL: NCT00651456
Title: A Phase II-III Randomized Trial Pemetrexed-Cisplatin Chemotherapy With or Without Bevacizumab (Avastin), 15 mg/kg, for Malignant Pleural Mesothelioma (MPM)
Brief Title: Mesothelioma Avastin Plus Pemetrexed-cisplatin Study
Acronym: MAPS
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Intergroupe Francophone de Cancerologie Thoracique (Other)
Collaborators: University Hospital, Caen (Other); Groupe Francais De Pneumo-Cancerologie (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IFCT-GFPC-0701
Record Dates: First submitted 2008-03-29; First posted 2008-04-02 (Estimated); Last update posted 2023-03-13 (Actual); Status verified 2023-03

CONDITIONS: Mesothelioma
MeSH Terms: conditions — Mesothelioma | interventions — Pemetrexed; Cisplatin; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Standard Chemotherapy
  Interventions: Drug: Standard Chemotherapy (Pemetrexed and Cisplatin)
- 2 (Experimental): Standard Chemotherapy + bevacizumab (Avastin)
  Interventions: Drug: Standard Chemotherapy (Pemetrexed and Cisplatin) + Bevacizumab

INTERVENTIONS:
Drug: Standard Chemotherapy (Pemetrexed and Cisplatin) — * Pemetrexed 500 mg/m² with previous Folic acid and vitamin B12 supplementation Day 1 (D1=D22, 6 cycles)
  * Cisplatin 75 mg/m² Day 1 (D1=D22, 6 cycles)
  Arms: 1
Drug: Standard Chemotherapy (Pemetrexed and Cisplatin) + Bevacizumab — * Pemetrexed 500 mg/m² with previous Folic acid and vitamin B12 supplementation D1 (D1=D22, 6 cycles)
  * Cisplatin 75 mg/m2 D1 (D1=D22, 6 cycles)
  * Bevacizumab 15 mg/kg D1 (D1=D22, until progression)
  Arms: 2

SUMMARY:
Our hypothesis is that the addition of bevacizumab to the standard chemotherapy treatment of MPM will improve overall survival and quality of life beyond that achieved with chemotherapy alone.

DETAILED DESCRIPTION:
A phase II trial associating the reference chemotherapy (pemetrexed plus cisplatin) with bevacizumab is needed to ensure that no specific toxicity is induced by this association, and that this triplet have interesting activity. As pleural mesothélioma is a rare tumor, a phase III trial, using the survival data from the phase II part study, will be able to include a sufficient number of patients, in a reasonable period of time, to answer the question of efficacy of the anti-angiogenic triplet, providing the efficacy outcomes could be considered as favorable, at the end of the phase II part of the study.

ELIGIBILITY:
Inclusion Criteria:

* Malignant, histologically proved, non resectable pleural Mesothelioma
* In case of pleural effusion, a talc pleurodesis, although not recommended, is allowed in accordance with current local practice, at the time of diagnostic thorascopy, with inclusion CT scan performed after pleurodesis.
* ECOG Performance status 0-2
* Mesothelioma with only pleural effusion without uni- or bidimensionally measurable disease will be eligible (adapted RECIST criteria)
* At least 18 years of age, less than 76 years of age
* Radiation therapy of thoracocentis tract (3 x 7Gy) performed before beginning medical study treatment, and the interval between thoracoscopic procedure and radiation will not exceed 28 days

Exclusion Criteria:

* Prior chemotherapy
* Brain metastasis
* History of cerebral vascular accident (CVA) or transient ischemic attack

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 448 (Actual)
Dates: Start 2008-02; Primary Completion 2015-01 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
% of patients with controled disease (responder and stable patients) at 6 months | 3-month

SECONDARY OUTCOMES:
Overall Survival | month
Number of participants with treatment-related adverse events as assessed by CTCAE v3.0 | month

OTHER OUTCOMES:
Medico-economic assessments of drugs (direct/indirect costs) | 3-month

CONTACTS AND LOCATIONS:
Overall Officials: Gilles Robinet, Dr, Study Director — GFPC; Arnaud Scherpereel, Dr, Study Director — Intergroupe Francophone de Cancerologie Thoracique
Locations (81):
- France (81):
  - Centre Hospitalier du Pays d'Aix, Aix-en-Provence
  - Annemasse - CH, Ambilly
  - Amiens - CHU, Amiens
  - Clinique de l'Europe, Amiens
  - Angers - CHU, Angers
  - Auxerre - CH, Auxerre
  - CHU Besancon - Pneumologie, Besançon
  - Béziers - CH, Béziers
  - Bobigny - Hôpital Avicenne, Bobigny
  - Bois-Guillaume - CHU, Bois-Guillaume
  - Boujan sur Libron - Polyclinique Saint-Privat, Boujan-sur-Libron
  - Hôpital Ambroise Paré - Pneumologie, Boulogne
  - Brest - CHU, Brest
  - Brest - HIA, Brest
  - Caen - Centre François Baclesse, Caen
  - CHU - Pneumologie, Caen
  - Chauny - CH, Chauny
  - Cherbourg - CH, Cherbourg
  - Hôpital Percy-Armées - Pneumologie, Clamart
  - CHU, Clermont-Ferrand
  - Colmar - CH, Colmar
  - Créteil - CHI, Créteil
  - Denain - CH, Denain
  - Centre Georges François Leclerc, Dijon
  - CHU Hôpital du Bocage, Dijon
  - Elbeuf - CH, Elbeuf
  - Evreux - CH, Évreux
  - Flers - CH, Flers
  - CHU Grenoble - pneumologie, Grenoble
  - Chartres - CH, Le Coudray
  - Centre Hospitalier - Pneumologie, Le Havre
  - Le Havre - HPE, Le Havre
  - Centre Hospitalier - Pneumologie, Le Mans
  - Le Mans - Clinique Victor Hugo, Le Mans
  - CHU (Hôpital Calmette) - Pneumologie, Lille
  - Limoges - Hôpital du Cluzeau, Limoges
  - CH de Longjumeau, Longjumeau
  - Lorient - CHBS, Lorient
  - Centre Léon Bérard, Lyon
  - HCL - Croix-Rousse, Lyon
  - APHM - Hôpital Sainte Marguerite, Marseille
  - Meaux - CH, Meaux
  - Mont de Marsan - CH, Mont-de-Marsan
  - Montpellier - CHRU, Montpellier
  - Mulhouse - CH, Mulhouse
  - CHU, Nancy
  - Nantes - Centre René Gauducheau, Nantes
  - Narbonne - Polyclinique Le Languedoc, Narbonne
  - Nevers - CH, Nevers
  - Nice - CAC, Nice
  - Orléans - CH, Orléans
  - Paray Le Monial - CH, Paray-le-Monial
  - Paray Le Monial - Clinique, Paray-le-Monial
  - Paris - Saint Louis, Paris
  - APHP - Hopital Tenon - Pneumologie, Paris
  - Paris - Curie, Paris
  - Pau - CH, Pau
  - HCL - Lyon Sud (Pneumologie), Pierre-Bénite
  - CHU, Poitiers
  - Pontoise - CH, Pontoise
  - Reims - CHU, Reims
  - Rennes - CHU, Rennes
  - Roubaix - CH, Roubaix
  - Rouen - CHU, Rouen
  - Saint Brieuc - CHG, Saint-Brieuc
  - Centre Etienne Dolet, Saint-Nazaire
  - Saint-Nazaire - CH, Saint-Nazaire
  - Institut de Cancérologie de la Loire, Saint-Priest-en-Jarez
  - Saint Quentin - CH, Saint-Quentin
  - Saint-Malo - CH, St-Malo
  - Strasbourg - NHC, Strasbourg
  - Suresnes - Hopital Foch, Suresnes
  - Thonon les bains - CH, Thonon-les-Bains
  - Toulon - CHI, Toulon
  - CHU Toulouse - Pneumologie, Toulouse
  - Tours - CHU, Tours
  - CH Valence, Valence
  - Valenciennes - Clinique, Valenciennes
  - CHI de la Haute-Saône - Pneumologie, Vesoul
  - CH de Villefranche - Pneumologie, Villefranche
  - Institut Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Zalcman G, Mazieres J, Margery J, Greillier L, Audigier-Valette C, Moro-Sibilot D, Molinier O, Corre R, Monnet I, Gounant V, Riviere F, Janicot H, Gervais R, Locher C, Milleron B, Tran Q, Lebitasy MP, Morin F, Creveuil C, Parienti JJ, Scherpereel A; French Cooperative Thoracic Intergroup (IFCT). Bevacizumab for newly diagnosed pleural mesothelioma in the Mesothelioma Avastin Cisplatin Pemetrexed Study (MAPS): a randomised, controlled, open-label, phase 3 trial. Lancet. 2016 Apr 2;387(10026):1405-1414. doi: 10.1016/S0140-6736(15)01238-6. Epub 2015 Dec 21. PMID 26719230
- [Derived] Levallet G, Dubois F, Elie N, Creveuil C, Brosseau S, Danel C, Scherpereel A, Lantuejoul S, Mazieres J, Greillier L, Audigier-Valette C, Bergot E, Moro-Sibilot D, Molinier O, Lena H, Monnet I, Morin F, Gounant V, Zalcman G. VEGFR2 and CD34 expression associated with longer survival in patients with pleural mesothelioma in the IFCT-GFPC-0701 MAPS phase 3 trial. Lung Cancer. 2023 Aug;182:107287. doi: 10.1016/j.lungcan.2023.107287. Epub 2023 Jun 26. PMID 37393757
- [Derived] Brosseau S, Danel C, Scherpereel A, Mazieres J, Lantuejoul S, Margery J, Greillier L, Audigier-Valette C, Gounant V, Antoine M, Moro-Sibilot D, Rouquette I, Molinier O, Corre R, Monnet I, Langlais A, Morin F, Bergot E, Zalcman G, Levallet G. Shorter Survival in Malignant Pleural Mesothelioma Patients With High PD-L1 Expression Associated With Sarcomatoid or Biphasic Histology Subtype: A Series of 214 Cases From the Bio-MAPS Cohort. Clin Lung Cancer. 2019 Sep;20(5):e564-e575. doi: 10.1016/j.cllc.2019.04.010. Epub 2019 May 13. PMID 31279641
- [Derived] Ribi K, Luo W, Colleoni M, Karlsson P, Chirgwin J, Aebi S, Jerusalem G, Neven P, Di Lauro V, Gomez HL, Ruhstaller T, Abdi E, Biganzoli L, Muller B, Barbeaux A, Graas MP, Rabaglio M, Francis PA, Foukakis T, Pagani O, Graiff C, Vorobiof D, Maibach R, Di Leo A, Gelber RD, Goldhirsch A, Coates AS, Regan MM, Bernhard J; SOLE Investigators. Quality of life under extended continuous versus intermittent adjuvant letrozole in lymph node-positive, early breast cancer patients: the SOLE randomised phase 3 trial. Br J Cancer. 2019 May;120(10):959-967. doi: 10.1038/s41416-019-0435-4. Epub 2019 Apr 10. PMID 30967649
- See also: Official website — http://www.ifct.fr